CLINICAL TRIAL: NCT03568591
Title: A Parallel-Group Controlled Trial Examining the Efficacy of a Psychosomatic Intervention
Brief Title: The Efficacy of a Psychosomatic Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff Metropolitan University (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Principal Investigator, Kirsty Hodgson, Principal Investigator - Research Lead, Cardiff Metropolitan University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LMT1131992C
Record Dates: First submitted 2018-05-21; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Type D Personality; Trauma, Psychological
Keywords: Psychosensory Therapy; Trauma, Psychological; DS14; CD-RISC; Resilience; Psychosomatic Medicine; Type D Personality; Salivary Cortisol; Blood Pressure; Havening Techniques
MeSH Terms: conditions — Psychological Trauma

STUDY DESIGN:
Intervention Model Description: A researcher-blind parallel-group controlled psychosomatic therapy intervention trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Coded-analysis group allocation and database - blind to allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Treatment) (Experimental): A treatment group cohort who have self-referred for the psychosensory therapy intervention (Havening Techniques).
  Interventions: Procedure: Psychosensory Therapy
- Control Group (Waiting List) (No Intervention): Self-referral waiting list cohort (usual care).

INTERVENTIONS:
Procedure: Psychosensory Therapy — Havening Techniques are a psychosensory therapy that incorporate the application of sensory input to alter neurochemical responses influencing thought, emotion and behaviour (Ruden, 2011).
  Other Names: Havening Techniques; Psychosomatic Intervention
  Arms: Intervention Group (Treatment)

SUMMARY:
This study examines the efficacy of a psychosensory intervention in relation to: Resilience, Type D personality, and physiological effects (on blood pressure, heart rate and salivary cortisol) in a group of people who have self-referred for the trauma resolution psychosensory therapy - Havening Techniques (HT).

DETAILED DESCRIPTION:
This study utilizes a single blind (researcher blind) comparison of the psychosensory therapy Havening Techniques (treatment) versus waiting list (no treatment). Participants will be assessed using resilience testing (CD-RISC), and Type D measure of personality (DS14). A subgroup of the treatment arm will be assessed for the biomarkers of blood pressure, heart rate and cortisol. This parallel-group controlled trial will examine the efficacy of Havening Techniques at 3 timepoints; baseline (Time point 1), twenty-four hours post (Time point 2) and one month later (Time point 3).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* Cognisant adults living in the United Kingdom.
* Will have self-referred for Havening Techniques trauma therapy.

Exclusion Criteria:

* Receiving any other therapeutic or pharmaceutical intervention in parallel.
* For the psychobiological evaluation subgroup: a history of HIV, Tuberculosis or Hepatitis B due to laboratory regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-06-11 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Change from the baseline DS14 measure of Type D personality scores at time point 2. | 24 hours post intervention (Time point 2) versus pre-intervention (Time point 1)
  Co-primary outcome measure: The DS14 measure of Type D personality is a 14-item questionnaire that uses a 5-point likert scale, each item weighted from 0 to 4. The DS14 incorporates the two 7-item subscales measuring the negative affect and social inhibition constituents of Type D personality (Denollet, 2005).
Change from the baseline Connor-Davidson Resilience Scale (CD-RISC) scores at time point 2. | 24 hours post intervention (Time point 2) versus pre-intervention (Time point 1)
  Co-primary outcome measure: The Connor-Davidson Resilience Scale (CD-RISC) assesses resilience and constitutes a 25=item questionnaire scored on a 5-point likert scale (rated 0-4). This scale has been successfully applied to evaluate change in intervention studies targeted at resilience (Connor and Davidson, 2003).

SECONDARY OUTCOMES:
Change in the DS14 measure of Type D personality score at time point 3. | 1 month post intervention (Time point 3)
  Repeat assessment of co-primary outcome measure 1.
Change in the Connor-Davidson Resilience Scale (CD-RISC) score at time point 3. | 1 month post intervention (Time point 3)
  Repeat assessment of co-primary outcome measure 2.
Change in Systolic Blood Pressure from baseline to time point 2. | 24 hours post intervention (Time point 2) versus pre-intervention (Time point 1)
  Systolic blood pressure will be assessed following rest in a sitting position (using an Omron hem 722c device).
Change in Systolic Blood Pressure at time point 3. | 1 month post intervention (Time point 3)
  Systolic blood pressure will be assessed following rest in a sitting position (using an Omron hem 722c device).
Change in Diastolic Blood Pressure from baseline to time point 2. | 24 hours post intervention (Time point 2) versus pre-intervention (Time point 1)
  Diastolic blood pressure and heart rate will be assessed following rest in a sitting position (using an Omron hem 722c device).
Change in Diastolic Blood Pressure at time point 3. | 1 month post intervention (Time point 3)
  Diastolic blood pressure and heart rate will be assessed following rest in a sitting position (using an Omron hem 722c device).
Change in Heart Rate from baseline to time point 2. | 24 hours post intervention (Time point 2) versus pre-intervention (Time point 1)
  Heart rate will be assessed following rest in a sitting position (using an Omron hem 722c device).
Change in Heart Rate at time point 3. | 1 month post intervention (Time point 3)
  Heart rate will be assessed following rest in a sitting position (using an Omron hem 722c device).
Change in Salivary Cortisol levels from baseline to time point 2. | 24 hours post intervention (Time point 2) versus pre-intervention (Time point 1)
  Salivette recordings taken at identical times of day (to avoid circadian influences) following rest in a sitting position. Dietary consistency and avoidance of alcohol advised to avoid confounding variables. Samples to be analysed by the clinical laboratory.
Change in Salivary Cortisol Levels at time point 3. | 1 month post intervention (Time point 3)
  Salivette recordings taken at identical times of day (to avoid circadian influences) following rest in a sitting position. Dietary consistency and avoidance of alcohol advised to avoid confounding variables. Samples to be analysed by the clinical laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Hodgson, Principal Investigator — Psychology Department, Cardiff Metropolitan University
Locations (1):
- Psychology Department, Cardiff, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Denollet J. DS14: standard assessment of negative affectivity, social inhibition, and Type D personality. Psychosom Med. 2005 Jan-Feb;67(1):89-97. doi: 10.1097/01.psy.0000149256.81953.49. PMID 15673629
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- See also: Ruden, R. (2011) When the Past is Always Present - Emotional Traumatisation, Causes, and Cures. USA: Routledge. — https://www.routledge.com/When-the-Past-Is-Always-Present-Emotional-Traumatization-Causes-and/Ruden/p/book/9780415875646